CLINICAL TRIAL: NCT01119430
Title: Fluoxetine Versus Fluoxetine Plus DU125530 in Latency of Antidepressant Response Shortening in Major Depressive Disorder
Brief Title: Fluoxetine Versus Fluoxetine Plus DU125530 in Major Depressive Disorder
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: interim analysis suggested no differences with whole sample
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSP-2003-01
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2010-05-07 (Estimated); Status verified 2010-05

CONDITIONS: Major Depression
Keywords: major depression; DU 125530; Treatment depression; Latency antidepressant
MeSH Terms: conditions — Depressive Disorder, Major | interventions — 1,2-benzisothiazol-3(2H)-one, 2-(4-(4-(7-chloro-2,3-dihydro-1,4-benzodioxin-5-yl)-1-piperazinyl)butyl)-, 1,1-dioxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluoxetine plus placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Fluoxetine plus DU125530 (Active Comparator)
  Interventions: Drug: DU125530

INTERVENTIONS:
Drug: DU125530 — 20mg/twice a day
  Other Names: Fluoxetine+DU
  Arms: Fluoxetine plus DU125530
Drug: Placebo — Similar pill as active comparator twice a day
  Other Names: Fluoxetine+placebo
  Arms: Fluoxetine plus placebo

SUMMARY:
The purpose of this study is to examine whether the speed of the clinical antidepressant action of fluoxetine can be accelerated by administering DU125530 a full 5-HT1A antagonist.

DETAILED DESCRIPTION:
SSRI acts by blocking the serotonin transporter (5-HT), increasing the availability of serotonin at the synaptic cleft averting its reuptake. The increment of serotonin activates 5-HT1A presynaptic autoreceptors, resulting in a modulation in the release of serotonin by the presynaptic neuron. It is proposed that 5-HT1A receptor antagonism could accelerate the clinical effect of antidepressants by preventing this negative feedback.Preclinical data obtained with selective 5-HT1A antagonists, such as pindolol, and with mice lacking 5-HT1a receptors supports this hypothesis. Results on partial antagonists (pindolol) are conclusive in accelerating SSRI. It is reasonable to call into question whether a total antagonism of 5-HT1a receptors could imply a more rapid antidepressant response. To test this hypothesis we conducted a double blind, randomised, controlled trial with DU 123550 added to fluoxetine 20 mg/day

ELIGIBILITY:
Inclusion Criteria:

* Consecutive eligible patients aged 18 to 70
* Diagnosis of unipolar major depression using DSM-IV criteria with moderate to severe symptoms (score e 18 on the Hamilton Depression Rating Scale-HDRS- of 17 items).
* There was a wash-out of 1 week of any antidepressant drug (specifically 28 days for fluoxetine) prior entering the study.
* Written informed consent was obtained from all participants.

Exclusion Criteria:

* Concurrent psychiatric disorders (DSM IV axis I, II cluster A or B)
* Failure to respond to drug treatment in current depressive episode
* Previous resistance to SSRIs or other antidepressant drug
* Suicide risk score e 3 on the HDRS.
* Participation in other drug trials within the previous month
* Presence of delusions or hallucinations
* History of substance abuse (including alcohol) in the past three months
* Pregnancy or lactation
* Organic brain disease or history of seizures
* Serious organic illnesses such as hypo or hyperthyroidism,cardiac arrhythmias, asthma, diabetes mellitus.
* Myocardial infarction in the past 6 month
* Frequent or severe allergic reactions
* Concomitant use of other psychotropic drugs (benzodiazepines were allowed), lockers or catecholamine-depleting agents
* Current structured psychotherapy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2004-05; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Scores on Hamilton Depression Rating Scale | 8 time points through 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Victor Pérez, MD, PhD, Principal Investigator — Psychiatrist, Hospital de Sant Pau; Enric Álvarez, MD, PhD, Principal Investigator — Head of Departement, Psiquiatria, Hospital de Sant Pau; Dolors Puigdemont, MD, Study Chair — Psychiatrist, Hospital de Sant Pau; Josefina Pérez, MD, Study Director — Psychiatrist, Hospital de Sant Pau
Locations (1):
- Hospital de Sant Pau, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Scorza MC, Llado-Pelfort L, Oller S, Cortes R, Puigdemont D, Portella MJ, Perez-Egea R, Alvarez E, Celada P, Perez V, Artigas F. Preclinical and clinical characterization of the selective 5-HT(1A) receptor antagonist DU-125530 for antidepressant treatment. Br J Pharmacol. 2012 Nov;167(5):1021-34. doi: 10.1111/j.1476-5381.2011.01770.x. PMID 22050051